CLINICAL TRIAL: NCT06979960
Title: The Effect of Face-to-Face and Online Training on Cancer Screening on Women's Knowledge, Attıtude and Shyness
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Melike Kutluol, principal investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/5731
Record Dates: First submitted 2025-05-02; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-02

CONDITIONS: Being Literate; Not Having Any Cognitive, Visual or Orthopedic Disabilities; Being Between the Ages of 50-65; Having a Smart Phone; The Effect of Education on Cancer Screening on the Knowledge Level of Women; The Effect of Education on Cancer Screening on Women&Amp;#39;s Attitudes; The Effect of Education on Cancer Screening on Women&Amp;#39;s Shyness Level
Keywords: cancer screenings; midwife; knowledge; attitude; shyness; woman; online education
MeSH Terms: conditions — Behavior; Shyness

STUDY DESIGN:
Intervention Model Description: Experimental Group; First interview: The women in the experimental group who applied to the Ketem unit were met and informed about the study. After the consent of the women who agreed to participate in the research was obtained; Personal information form and scales were applied. Then the first part of the training session was held. For the second phase of the training session, the appointment place, day and time were determined one week later. Participants were given a training booklet. Second meeting: In the second meeting, 1 week after the first training, the second part of the training, namely breast cancer screening program, cervical cancer screening program and colorectal cancer screening program, was held.Third interview: A reminder training was held over the phone 1 weekafter the second training.Fourth interview: Post-test data were obtained by telephone by the researcher 2 weeks after the reminder training was implemented.Control Group;no action taken
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training group (Experimental): First interview: The women in the experimental group who applied to the Ketem unit were met and informed about the study. After the consent of the women who agreed to participate in the research was obtained; Personal information form and scales were applied. Then the first part of the training session was held. For the second phase of the training session, the appointment place, day and time were determined one week later. Participants were given a training booklet.
  Second meeting: In the second meeting, 1 week after the first training, the second part of the training, namely breast cancer screening program, cervical cancer screening program and colorectal cancer screening program, was held.
  Third interview: A reminder training was held over the phone 1 week after the second training.
  Fourth interview: Post-test data were obtained by telephone by the researcher 2 weeks after the reminder training was implemented.
  Interventions: Behavioral: cancer screening education
- control group (No Intervention): The women in the control group who applied to the Ketem unit were introduced to the first interview and their written consent was obtained, and then the personal information form and scales were applied. After the personal information form and scales were applied again 4 weeks after the first interview, the post-test data were obtained. After the post-test data were obtained, the women in the control group, who were not subjected to any intervention, were given an educational booklet in line with the "Equality" principle.

INTERVENTIONS:
Behavioral: cancer screening education — It will be carried out to examine the effect of the educational intervention given using the cancer screening training booklet on women's knowledge, attitude and shyness levels.
  Arms: training group

SUMMARY:
Cancer is a large group of diseases that occur due to abnormal cell proliferation in almost all organs of the body. Cancer is the second leading cause of death in the world after cardiovascular diseases. The fact that cancer is a preventable disease reveals the importance of cancer screenings. Cancer screening aims to detect it in the early stages when the chance of treatment is high. Screening programs for breast cancer, cervical cancer and colorectal cancer are recommended by WHO. In order for these screening programs to achieve their goals, people within the scope of screening must participate in screening. However, there are many factors involved in participating in these screening programs. Even though health professionals direct people to screening programs, at this point people's knowledge, attitude and shyness levels affect their participation in screening programs. The research is planned to be experimentally pre-test-post-test, and the data will be collected before and after the training to be given face-to-face and online by the researcher. The results obtained as a result of the study will be taken into consideration by midwives in terms of the effect of the education given on cancer screenings on women's knowledge, attitude and shyness levels.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 50-65
* Being literate
* Having a smart mobile phone
* No cognitive, visual or orthopedic disabilities

Exclusion Criteria:

* Not answering questions completely. Being diagnosed with a psychiatric disease.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 68 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Knowledge Scale for Cancer Screening | first day encountered
  This scale, which consists of 25 items and 3 sub-dimensions, has no special names for its sub-dimensions. The scale; The items in the 1st sub-dimension are items 8, 17-23, 25, 28, totaling 10 items, The items in the 2nd sub-dimension are items 4, 5, 7, 10, 12,13, 15, 16, 27, totaling 9 items,The items in the 3rd sub-dimension are items 1-3, 9, 11, 24, totaling 6 items. This scale, which is answered in a range from 1 to 3 as ''1: True, 2: False, 3: I don't know'', is a three-point rating type. When calculating the scale score, the ''True'' answers are given 1 point, and the ''False'' and ''I don't know'' answers are given 0 points. The lowest possible score for this scale is 0, and the highest possible score is 25. Items 2, 11, and 24 of this scale, which has three negatively connoted items, should be reverse coded. The order of use of the items in the scale is not important and researchers can use them in a mixed order.
Attitude Scale Towards Cancer Screening | first day encountered
  The Attitude Scale Towards Cancer Screenings was developed by Yıldırım Öztürk and his colleagues in 2020, and its Turkish validity and reliability study was conducted. This scale, consisting of 24 items and a single dimension, is a five-point Likert-type scale. The items of the scale, which are answered in the range of 1 to 5, are as follows: 1: I completely disagree, 2: I somewhat disagree, 3: I neither agree nor disagree, 4: I somewhat agree, 5: I completely agree. This scale is suitable for evaluating individuals whose age range is 30-70, whose education level is at least literate, and who do not have cognitive, visual or orthopedic disabilities that would prevent them from answering the questions on the scale. There is no specific cut-off point for this scale, where the lowest score is 24 and the highest is 120.Scores close to 24 on the scale indicate that individuals have a negative attitude towards cancer screening.
Shyness scale | first day encountered
  This scale, which is a 5-point Likert-type scale ranging from 1 to 5, has 20 items that include expressions regarding feelings and behaviors that can be used to determine how shy individuals perceive themselves as. Individuals are asked to mark one of the following answers opposite the statements on the scale: "Not at all suitable for me," "Not suitable," "Undecided," or "Very suitable for me." As a result, the calculation is made by giving 1 (One) point to the item "Not at all suitable for me," 2 (Two) points to the item "Not suitable for me," 3 (Three) points to the item "Undecided," 4 (Four) points to the item "Suitable for me," and 5 (Five) points to the item "Very suitable for me." The lowest score that can be obtained from the scale is 20, while the highest score is 100. A high score on the scale indicates that the individual perceives himself as "shy."

SECONDARY OUTCOMES:
Attitude Scale Towards Cancer Screening | up to 4th week after registration
  The Attitude Scale Towards Cancer Screenings was developed by Yıldırım Öztürk and his colleagues in 2020, and its Turkish validity and reliability study was conducted. This scale, consisting of 24 items and a single dimension, is a five-point Likert-type scale. The items of the scale, which are answered in the range of 1 to 5, are as follows: 1: I completely disagree, 2: I somewhat disagree, 3: I neither agree nor disagree, 4: I somewhat agree, 5: I completely agree. This scale is suitable for evaluating individuals whose age range is 30-70, whose education level is at least literate, and who do not have cognitive, visual or orthopedic disabilities that would prevent them from answering the questions on the scale. There is no specific cut-off point for this scale, where the lowest score is 24 and the highest is 120. Scores close to 24 on the scale indicate that individuals have a negative attitude towards cancer screening.
Knowledge Scale for Cancer Screening | up to 4th week after registration
  This scale, which consists of 25 items and 3 sub-dimensions, has no special names for its sub-dimensions. The scale; The items in the 1st sub-dimension are items 8, 17-23, 25, 28, totaling 10 items, The items in the 2nd sub-dimension are items 4, 5, 7, 10, 12,13, 15, 16, 27, totaling 9 items,The items in the 3rd sub-dimension are items 1-3, 9, 11, 24, totaling 6 items. This scale, which is answered in a range from 1 to 3 as ''1: True, 2: False, 3: I don't know'', is a three-point rating type. When calculating the scale score, the ''True'' answers are given 1 point, and the ''False'' and ''I don't know'' answers are given 0 points. The lowest possible score for this scale is 0, and the highest possible score is 25. Items 2, 11, and 24 of this scale, which has three negatively connoted items, should be reverse coded. The order of use of the items in the scale is not important and researchers can use them in a mixed order.
Shyness scale | up to 4th week after registration
  This scale, which is a 5-point Likert-type scale ranging from 1 to 5, has 20 items that include expressions regarding feelings and behaviors that can be used to determine how shy individuals perceive themselves as. Individuals are asked to mark one of the following answers opposite the statements on the scale: "Not at all suitable for me," "Not suitable," "Undecided," or "Very suitable for me." As a result, the calculation is made by giving 1 (One) point to the item "Not at all suitable for me," 2 (Two) points to the item "Not suitable for me," 3 (Three) points to the item "Undecided," 4 (Four) points to the item "Suitable for me," and 5 (Five) points to the item "Very suitable for me." The lowest score that can be obtained from the scale is 20, while the highest score is 100. A high score on the scale indicates that the individual perceives himself as "shy."

CONTACTS AND LOCATIONS:
Locations (1):
- Inönü University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD underlying results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR